CLINICAL TRIAL: NCT05642910
Title: The Efficacy of Azvudine and Paxlovid in High-risk Patients With COVID-19: A Prospective Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Collaborators: Hohhot First Hospital, Hohhot, Inner Mongolia, China (Unknown)
Responsible Party: Principal Investigator, Songqiao Liu, MD. PhD., Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBR2022072
Record Dates: First submitted 2022-12-07; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: SARS-CoV-2 Infection
Keywords: SARS-CoV-2; antivirus; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — azvudine; Control Groups

STUDY DESIGN:
Intervention Model Description: Patients who meet inclusion criteria will be randomized into the Azvudine group (treatment group) and Paxlovid group (control group).
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azvudine group (Experimental): Patients received Azvudine orally, for 7 consecutive days (7 doses in total) .
  Interventions: Drug: Azvudine
- Paxlovid group (Active Comparator): Patients received Paxlovid orally for 5 consecutive days (10 doses in total).
  Interventions: Drug: Paxlovid group

INTERVENTIONS:
Drug: Azvudine — Patients received Azvudine orally, for 7 consecutive days (7 doses in total)
  Other Names: treatment group
  Arms: Azvudine group
Drug: Paxlovid group — Patients received Paxlovid orally for 5 consecutive days (10 doses in total).
  Other Names: control group
  Arms: Paxlovid group

SUMMARY:
This is a randomized controlled clinical study on the clinical efficacy of Azvudine and Paxlovid antivirus therapy in COVID-19 patients with high-risk. The objective is to examine the effect of high-risk on the time for COVID-19 patients to achieve 2 continuously negative SARS-CoV-2 nucleic acid test result, and the RT-PCR negative conversion rates in day 7. Patients who meet inclusion criteria will be randomized into the Azvudine group (treatment group) and Paxlovid group (control group).

DETAILED DESCRIPTION:
After enrollment, patients will be randomized into treatment or control groups. Patients received Azvudine orally, for 7 consecutive days (7 doses in total) or Paxlovid orally for 5 consecutive days (10 doses in total). The test for RT-PCR test through either nasopharyngeal or oropharyngeal swabs were conducted on a daily basis from day 3 of their hospitalization until conversion was observed. The primary outcome was the proportion of patients acheive 2 continuously RT-PCR negative for SARS-CoV-2 at 7 days following treatment initiation, including both ORF gene Ct value≥35 and N gene Ct value≥35. Secondary outcomes included 1) the proportion of patients RT-PCR negative for SARS-CoV-2 at 14 days; 2) the time to conversion from a positive RT-PCR test to 2 continuously negative test; 3) 14-day treatment failure rate (need mechanical ventilation or high-flow oxygen therapy or death).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85 years (inclusive).
* Meet the diagnostic criteria for COVID-19.
* At least one high risk factor for progression to severe COVID-19
* No more than 5 days from the onset of clinical symptoms
* Sign informed consent form.

Exclusion Criteria:

* Severe or critically patients with COVID-19
* Have received neutralizing antibodies or convalescent plasma therapy due to COVID-19
* Child-Pugh grade C or acute liver failure
* Chronic renal failure (eGFR<30 mL/min)
* Grade III or IV cardiac function, or known left ventricular ejection fraction < 30%
* Known or suspected history of active or extrapulmonary tuberculosis
* Patients who are allergic to the active ingredient of the drug
* Pregnant and lactating women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients RT-PCR negative for SARS-CoV-2 at 7 days | 7 days after enrolled
  the proportion of patients RT-PCR negative for SARS-CoV-2 at 7 days

SECONDARY OUTCOMES:
the proportion of patients RT-PCR negative for SARS-CoV-2 at 14 days | 14 days
  the proportion of patients RT-PCR negative for SARS-CoV-2 at 14 days
the time to conversion from a positive RT-PCR test to 2 continuously negative test | 14 days
  the time to conversion from a positive RT-PCR test to 2 continuously negative test

CONTACTS AND LOCATIONS:
Overall Officials: Songqiao Liu, MD. PhD., Principal Investigator — Southeast university
Locations (1):
- Hohhot First Hospital, Hohhot, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: No
We did not seek or receive approval for this data sharing from our Institutional Review Board .